CLINICAL TRIAL: NCT00282646
Title: (Intraarterial Progenitor Cell Transplantation of Bone Marrow Mononuclear Cells for Induction of Neovascularization in Patients With Peripheral Arterial Occlusive Disease)
Brief Title: Safety and Feasibility Study of Autologous Bone Marrow Cell Transplantation in Patients With Peripheral Arterial Occlusive Disease (PAOD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, A. M. Zeiher, Prof. Dr. A.M. Zeiher, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-000968-33; PROVASA
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Arterial Occlusive Diseases
Keywords: critical limb ischemia; peripheral arterial occlusive disease; [C14.907.137]
MeSH Terms: conditions — Arterial Occlusive Diseases; Chronic Limb-Threatening Ischemia; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Intervention Model Description: Intraarterial administration of BM-MNC or placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): intraarterial application of bone marrow mononuclear cells
  Interventions: Procedure: intraarterial stem cell therapy; Other: Stem cells
- 2 (Placebo Comparator): intraarterial application of placebo
  Interventions: Procedure: intraarterial stem cell therapy; Other: Stem cells

INTERVENTIONS:
Procedure: intraarterial stem cell therapy — catheter delivery of stem cells
Other: Stem cells — intraarterial application of bone marrow mononuclear cells versus placebo

SUMMARY:
Patients with peripheral artery disease, stage III or IV who are not candidates for interventional or operative therapy should be treated with intraarterial progenitor cell therapy (autologous bone marrow cells) in a randomized, placebo controlled trial.

DETAILED DESCRIPTION:
Main goal:

Improvement of limb perfusion (Ankle brachial index).

Secondary aims:

Reduction of pain Reduction of Ulcer size Walking distance Improvement in tissue oxygenation (TCO2) Minor or major amputation

ELIGIBILITY:
Inclusion Criteria:

* Patients with PAOD (Stage III or IV)
* Distal arterial occlusions
* Patients with Buergers Disease
* Signed informed consent

Exclusion Criteria:

* Successful bypass operation or intervention within the last 3 months
* Active infection, feber, chronic inflammatory disease
* HIV, Hepatitis
* Tumor within the last 5 years, complete remission required
* Stroke or myocardial infarction within last 3 months
* Renal insufficiency (creatinine > 2 mg/dl)
* Liver disease (GOT > 2x upper limit oder spontaneous INR > 1,5).
* Anemia (hemoglobin < <10 mg/dl)
* Thrombocytopenia < 100.000/µl
* Allergies to Aspirin, Clopidogrel, Heparin
* Bleeding disorder
* Gastrointestinal bleeding within last 3 months
* Surgery or trauma within the last 2 months
* Pregnancy
* Mental retardation
* Inclusion in other clinical study within last 30 days

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-10; Primary Completion 2010-10 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Ankle brachial index | 6 months

SECONDARY OUTCOMES:
Ulcer size | 6 months
Pain | 6 months
Walking distance | 6 months
TCO2 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas M Zeiher, MD, Principal Investigator — Div. of Cardiology, University of Frankfurt, Germany; Dirk H Walter, MD, Study Director — Div. of Cardiology, University of Frankfurt, Germany
Locations (1):
- Div. of Cardiology and Vascular Medicine, Frankfurt, Germany

REFERENCES:
- [Derived] Sciahbasi A, Romagnoli E, Trani C, Burzotta F, Sarandrea A, Summaria F, Patrizi R, Rao S, Lioy E. Operator radiation exposure during percutaneous coronary procedures through the left or right radial approach: the TALENT dosimetric substudy. Circ Cardiovasc Interv. 2011 Jun;4(3):226-31. doi: 10.1161/CIRCINTERVENTIONS.111.961185. Epub 2011 May 17. PMID 21586692
- [Derived] Walter DH, Krankenberg H, Balzer JO, Kalka C, Baumgartner I, Schluter M, Tonn T, Seeger F, Dimmeler S, Lindhoff-Last E, Zeiher AM; PROVASA Investigators. Intraarterial administration of bone marrow mononuclear cells in patients with critical limb ischemia: a randomized-start, placebo-controlled pilot trial (PROVASA). Circ Cardiovasc Interv. 2011 Feb 1;4(1):26-37. doi: 10.1161/CIRCINTERVENTIONS.110.958348. Epub 2011 Jan 4. PMID 21205939